CLINICAL TRIAL: NCT03618589
Title: Comparison of Effectiveness of Opioid Only and Pregabalin add-on for the Treatment of Neuropathic Pain in Cervical Myelopathy Patients
Brief Title: Pregabalin add-on for Neuropathic Pain in Cervical Myelopathy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chun Kee Chung, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pregabalin & LANSS
Record Dates: First submitted 2018-07-09; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Pain, Neuropathic
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid only (Placebo Comparator): Patients in the opioid group received the only opioid (5mg of oxycodone three times a day) for 8 weeks.
  Interventions: Drug: Opioid
- pregabalin add-on (Experimental): Patients in the pregabalin add-on group received 75mg of pregabalin twice a day for the first week (150 mg/day) and 150mg of pregabalin twice a day (300 mg/day) for the second week and 300mg of pregabalin twice a day (600mg/day) for subsequent 6 weeks.
  Interventions: Drug: Pregabalin; Drug: Opioid

INTERVENTIONS:
Drug: Pregabalin — Patients in the pregabalin add-on group received 75mg of pregabalin twice a day for the first week (150 mg/day) and 150mg of pregabalin twice a day (300 mg/day) for the second week and 300mg of pregabalin twice a day (600mg/day) for subsequent 6 weeks.
  Other Names: Lyrica
  Arms: pregabalin add-on
Drug: Opioid — Patients in the opioid group received the only opioid (5mg of oxycodone three times a day) for 8 weeks.
  Other Names: IRcordon

SUMMARY:
There is no information on the effect of pregabalin in patients with neuropathic pain in cervical myelopathy under routine clinical practice.

The investigators will conduct this prospective, randomized trial to determine the efficacy of pregabalin for neuropathic pain in cervical myelopathic patients in order to validate or refute this popular practice. The primary aim of this study was to compare Leeds assessment of neuropathic symptoms and signs scale (LANSS) scores of neuropathic pain in cervical myelopathy patients.

DETAILED DESCRIPTION:
Neuropathic pain is a well-recognized clinical entity. It is defined as pain caused by the lesion or dysfunction of the peripheral or central nervous system, and it can be diagnosed by well-established clinical criteria. Neuropathic pain is caused by lesions or dysfunction of the nervous system and is initiated by several cellular and molecular mechanisms. Compression of neural and neurovascular structures may result in neuropathic pain. Although a number of therapies are available for neuropathic pain, including antidepressants, tramadol, opioids, and different antiepileptic drugs, the results of a recent systematic review suggest that, in view of their balance between efficacy and tolerability, pregabalin can be regarded as first line treatments for peripheral pain with a neuropathic component.

Pregabalin is one of antiepileptic drugs (AEDs) that have been studied in the treatment of a wide variety of disorders, such as neuropathic pain, epilepsy, spasticity, and anxiety. The use of AEDs in the treatment of neuropathic pain is based on a number of similarities in the pathophysiologic and biochemical mechanisms underlying neuropathic pain and epilepsy. Its use for the treatment of several neuropathic pain syndromes is common, and it is approved by the Food and Drug Administration (FDA) for the treatment of diabetic neuropathy, post-herpetic neuralgia, fibromyalgia and spinal cord injury, a model of central neuropathic pain. The off-label use of pregabalin for the various pain syndromes in general, and for neuropathic pain in particular, is ubiquitous. However, minimal support for this practice exists in the literature and its cost is perhaps exorbitant. There is no information on the effect of pregabalin in patients with neuropathic pain in cervical myelopathy under routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18 to 80 years
2. Among patients with cervical myelopathy, patients with neuropathic pain (LANSS pain scale ≥ 12)
3. Completing 8-week drug trial

Exclusion Criteria:

1. Current or prior gabapentin or pregabalin use
2. Chronic use of narcotic pain medications
3. Chronic depression or the use of anti-depressants
4. History of addiction and/or substance abuse
5. Presence of significant motor deficits, and /or bowel and/or bladder dysfunction
6. Known renal insufciency, diabetes, congestive heart failure, cardiac conduction abnormalities, and thrombocytopenia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11-26 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Leeds assessment of neuropathic symptoms and signs (LANSS) and visual analogue scale (VAS) | 2 months
  The LANSS pain scales are used globally to screen for the presence of pain of neuropathic origin because they have high sensitivity and specificity compared with other available tools. It rages from 0 to 24. The LANSS scores ≧12 suggest the presence of neuropathic pain.
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. It ranges from 0 to 10 (0 means no pain, 10 means worst pain.

SECONDARY OUTCOMES:
neck disability index (NDI) and EuroQol- 5 Dimension (EQ-5D) | 2 months
  The NDI is a modification of the Oswestry Low Back Pain Disability Index. It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. It ranges from 0 to 45 (0 means no disability, 45 means severe disability).
  The EQ-5D is a generic, self-completed, easy-to-use questionnaire. The EQ-5D comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). There are potentially 243 (=35) different health states.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Kee Chung, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No